CLINICAL TRIAL: NCT04016935
Title: EndoPredict® Extended Endocrine Trial (EXET): A Prospective Registry to Evaluate the Impact of EndoPredict® Test on Extended Endocrine Treatment Decisions and Patient Outcomes.
Brief Title: EndoPredict® Extended Endocrine Trial (EXET)
Status: Terminated | Type: Observational
Why Stopped: It was determined that we had sufficient enrollment and study data to explore the impact of the Endopredict test in endocrine therapy decision-making.
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC-010
Record Dates: First submitted 2019-06-26; First posted 2019-07-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Primary Invasive Breast Cancer
Keywords: ER+ and HER2- Breast Cancer patients; Extended Endocrine Therapy; EndoPredict; Additional Relevant MeSH terms:; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases
MeSH Terms: conditions — Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary invasive ER+ HER2- breast cancer: Distant recurrence-free survival (DRFS) between years 5 and 10 post-diagnosis of women with ER+, HER2- breast cancer who are classified as low risk according to their EPclin score and who did not receive extended endocrine therapy
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The purpose of this study is to evaluate the impact of using EndoPredict® clinically to inform treatment decisions for extended endocrine therapy, and the subsequent impact on patient outcomes.

DETAILED DESCRIPTION:
The EndoPredict® molecular test is validated to predict late distant recurrence after 5 years of endocrine therapy in women with estrogen receptor-positive (ER+), human epidermal growth factor receptor 2-negative (HER2-) early stage breast cancer, with or without treatment with adjuvant chemotherapy. The test provides an individualized EPclin score based on the tumor gene expression, tumor size and nodal status, and categorizes patients as High or Low risk of distant recurrence.

The primary objective of this study is to evaluate the distant recurrence-free survival (DRFS) at 5-10 years in patients with ER+/HER2- early stage breast cancer with EPclin Low scores that did not extend endocrine therapy.

Data collection is prospective and patient enrollment is expected to occur over 24 months. The study will enroll patients who are near the 5-year post-diagnosis time point when decisions on extending endocrine therapy are being made. Patient breast cancer tumors, stored from surgical collection after initial diagnosis, will be tested with EndoPredict and a report generated. The provider will convey the report results to the patient and establish a treatment plan to continue or forgo endocrine therapy. Patients will then be followed for 6 years with data collection every year, and outcomes (distant and local disease recurrence, second primary breast cancer, etc.) recorded.

The associations between outcomes and treatment, EPclin score and risk category, EP molecular score, and clinicopathologic features will be investigated in all patients and in subpopulations (node negative, node positive, treated with or without chemotherapy, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least 18 years of age at time of enrollment
* Able to provide informed consent
* ER+, HER2- breast tumor
* Stage T1-T3
* Currently receiving endocrine therapy
* Are between 4 and 6.5 years post-invasive breast cancer diagnosis
* Have all available information to produce an EPclin score, including treatment-naïve tumor stage, nodal status, and sufficient amount of remaining tissue from biopsy or resection to perform genomic testing (section 9)
* Patient and physician are willing to consider a change in endocrine therapy

Exclusion Criteria:

* Metastatic disease or currently active additional cancer diagnosis (except non- melanoma skin cancer) or any second primary breast cancer (includes ductal and/or lobular carcinoma in situ)
* Patient received systemic chemotherapy within 1 year of enrollment
* Currently enrolled in an interventional clinical trial or other clinical trial that precludes freely making decisions regarding extended endocrine therapy
* More than 3 positive nodes
* Received neo-adjuvant treatment (new-adjuvant chemotherapy or neo-adjuvant endocrine therapy)
* Are beyond 7 years post-breast cancer diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The primary objective of this study is to evaluate distant recurrence-free survival (DRFS) between years 5 and 10 post-diagnosis of women with ER+, HER2- breast cancer who are classified as low risk according to their EPclin score and who did not receive extended endocrine therapy.
Study Population: Approximately 2,800 patients with ER+, HER2- breast cancer will be enrolled in this study across multiple sites. These patients will include both node-positive and node negative patients, with a minimum of 1673 patients with low-risk EPclin scores including 1,505 who forego extended endocrine therapy. Patients will be eligible for the study if they meet the following inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 855 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluate DRFS of women 5-10 years post diagnosis with ER+, HER2-breast cancer who are low risk according to their EPclin scores | 10 Years
  The primary objective of this study is to evaluate distant recurrence-free survival (DRFS) between years 5 and 10 post-diagnosis of women with ER+, HER2- breast cancer who are classified as low risk according to their EPclin score and who did not receive extended endocrine therapy

SECONDARY OUTCOMES:
Evaluate DRFS between years 5 and 10 post-diagnosis in women classified as low risk according to their EPclin who received extended endocrine therapy | 10 Years
  Evaluate DRFS between years 5 and 10 post-diagnosis in women classified as low risk according to their EPclin who received extended endocrine therapy
Evaluate DRFS between years 5 and 10 post-diagnosis in women classified as high risk according to their EPclin score based on treatment decisions. | 10 Years
  Evaluate DRFS between years 5 and 10 post-diagnosis in women classified as high risk according to their EPclin score based on treatment decisions.
Evaluate adherence to EndoPredict® test results when making decisions regarding extended endocrine therapy | 1 Year
  Evaluate the proportion of patients classified as EPclin low who forgo extending endocrine and the proportion of EPclin high who extend endocrine therapy beyond 5 years
Evaluate adherence to EndoPredict® test results when making decisions regarding extended endocrine therapy according to whether patients received adjuvant chemotherapy. | 1 Year
  Evaluate the proportion of patients who received adjuvant chemotherapy classified as EPclin low who forgo extending endocrine and those classified as EPclin high who extend endocrine therapy beyond 5 years
Evaluate disease-free survival in patients stratified based on EPclin risk classification and actual treatment. | 10 Years
  Evaluate disease-free survival in patients stratified based on EPclin risk classification and actual treatment.

OTHER OUTCOMES:
Compare previous chemotherapy treatment decisions to chemotherapy treatment recommendations based on EndoPredict® risk classification. | 1 Year
  Compare previous chemotherapy treatment decisions to chemotherapy treatment recommendations based on EndoPredict® risk classification.
Repeat all primary and secondary objectives in subsets of patients based on variables such as clinicopathologic features and treatment. | 10 Years
  Repeat all primary and secondary objectives in subsets of patients based on variables such as clinicopathologic features and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaunessey, MD, Principal Investigator — US Oncology
Locations (51):
- United States (51):
  - Providence, Burbank, California
  - Sutter Hematology and Oncology, Roseville, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - AON Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - New York Oncology Hematology, Albany, New York
  - New York Oncology Hematology, Clifton Park, New York
  - Hematology Oncology Associates of Central New York, PC, East Syracuse, New York
  - Akron General Medical Center, Akron, Ohio
  - Summa Health, Akron, Ohio
  - UPMC Hillman Cancer Center Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center Upper St. Clair, Bethel Park, Pennsylvania
  - Butler Health System Medical Oncology, Butler, Pennsylvania
  - UPMC Hillman Cancer Center - Moon, Coraopolis, Pennsylvania
  - UPMC Passavant North Cranberry (OHA), Cranberry Township, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hillman Cancer Center Horizon, Farrell, Pennsylvania
  - UPMC Hillman Cancer Center Greenville, Greenville, Pennsylvania
  - UPMC Hillman Cancer Center Indiana, Indiana, Pennsylvania
  - UPMC Hillman Cancer Center Arnold Palmer at Norwin, Irwin, Pennsylvania
  - UPMC Hillman Cancer Center Murtha, Johnstown, Pennsylvania
  - UPMC Hillman Cancer McKeesport, McKeesport, Pennsylvania
  - Ortenzio Cancer Center, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center Arnold Palmer at Mt. Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Hillman Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center New Castle, New Castle, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center St Margaret, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Passavant (HOA), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Passavant (OHA), Pittsburgh, Pennsylvania
  - UPMC - St. Clair Hospital - Integrated Cancer Services, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Northwest, Seneca, Pennsylvania
  - UPMC Hillman Cancer Center Uniontown, Uniontown, Pennsylvania
  - UPMC Hillman Cancer Center Washington, Washington, Pennsylvania
  - UPMC Hillman Cancer Center Jefferson, West Mifflin, Pennsylvania
  - UPMC Hillman Cancer Center Williamsport, Williamsport, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Carolina Blood and Cancer Care Associates, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Hope Cancer of Texas, Tyler, Texas
  - Texas Oncology, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No